CLINICAL TRIAL: NCT07218523
Title: A Phase 3, Multicentre, Randomised (1:1), Parallel-group, Active-controlled, Central Reader Colonoscopist-blind Study to Evaluate the Bowel Cleansing Efficacy, Safety, Tolerability, Palatability, and Acceptability of PLENVU® as Compared to Sodium Picosulfate in Paediatric Participants From 1 to < 18 Years of Age in Preparation for Colonoscopy (CLARITY)
Brief Title: A Study to Investigate Bowel Cleansing With PLENVU® Compared to Sodium Picosulfate in Participants Aged 1 to < 18 Years of Age in Preparation for Colonoscopy
Acronym: CLARITY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NER1006-01/2025; 2025-522046-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Bowel Cleansing Prior to Clinical Procedures
Keywords: Colonoscopy; Paediatric; Harefield Cleansing Scale; Boston Bowel Preparation Scale; Plenvu; Polyethylene Glycol (PEG); Bowel Cleansing
MeSH Terms: interventions — Polyethylene Glycols; picosulfate sodium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The central reader colonoscopist will be blinded to the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLENVU® (Experimental): Participants will receive PLENVU® in a 2-day split dosing regimen.
  Interventions: Drug: PLENVU®
- Sodium picosulfate (Active Comparator): Participants will receive sodium picosulfate in a 2-day split dosing regimen according to the local label.
  Interventions: Drug: Sodium picosulfate

INTERVENTIONS:
Drug: PLENVU® — PLENVU® will be administered as an oral solution.
  Other Names: NER1006
  Arms: PLENVU®
Drug: Sodium picosulfate — Sodium picosulfate will be administered as an oral solution.
  Other Names: PICOPREP®; PICOLAX®
  Arms: Sodium picosulfate

SUMMARY:
The purpose of the study is to assess the efficacy, safety and tolerability of PLENVU® by measuring its bowel cleansing success rate compared to sodium picosulfate in paediatric participants aged less than 18 years who are scheduled to undergo a colonoscopy. Colonoscopy is a crucial procedure that helps to diagnose and manage various gastrointestinal (GI) conditions in paediatric patients. An adequate level of bowel preparation and cleansing is essential for effective colonoscopy to allow proper visualisation of the bowel.

DETAILED DESCRIPTION:
This is a multicentre, active-controlled study in which the participants will be randomised 1:1 into one of two treatment groups - PLENVU® or sodium picosulfate in a 2-day split dosing regimen. The study will include -

1. A Screening Period of up to 28 days (Day -28 to Day -1).
2. A Treatment Period (Day 1 to Day 2) - Participants will be randomised to receive either PLENVU® or sodium picosulfate. Participants will be admitted into the Clinical Research Unit (CRU) on Day 1 and will remain in the CRU for the duration of study intervention administration (Day 1 and Day 2) and colonoscopy (Day 2). Participants will be discharged on Day 2 following the colonoscopy and evaluation of colon cleansing.
3. A safety follow-up call or CRU visit (Day 9 ± 2 days).

ELIGIBILITY:
Inclusion Criteria:

* Participants who require a colonoscopy.
* Must weigh a minimum of 10 kg, and participants aged 1 to < 4 years of age must be above the 10th percentile of weight for age.
* Must have a negative urine pregnancy test (or serum if a urine pregnancy test cannot be confirmed as negative [e.g. three ambiguous results]) within 24 hours before the first dose of study intervention.
* Must use a highly effective method of contraception (failure rate < 1% per year) from Day 1 and throughout the Safety Follow-up Period.
* Must not be breastfeeding.
* Participant is able to receive regular external feeding without breastfeeding.

Exclusion Criteria:

* Has a past history within last 12 months or current episode of severe constipation (requiring repeated use of laxatives/enema or physical intervention before resolution).
* Has known or suspected ileus, GI obstruction, gastric retention, bowel perforation, toxic colitis, ischaemic colitis, or megacolon.
* Has ongoing severe acute inflammatory bowel disease that contraindicates colonoscopy.
* Participant has history of significant GI surgeries.
* Has known glucose-6-phosphate dehydrogenase (G6PD) deficiency or phenylketonuria.
* Participant has a past history within the last 12 months or evidence of any ongoing clinically relevant electrocardiogram (ECG) abnormalities (e.g. arrhythmias).
* Has a history of uncontrolled hypertension.
* Participant has regularly used laxatives or colon motility altering drugs in the last month (i.e. more than two times per week) and/or has used one or more laxatives within 72 hours prior to administration of the preparation.
* Has known hypersensitivity or allergic reaction to PEG, ascorbic acid, sodium picosulfate, magnesium oxide, or any other component of the investigational product or comparator.
* Received or scheduled to receive any vaccines or devices within one week prior to first dose of study intervention.
* Has a significant neurological disorder or a past history of seizures (excluding simple febrile seizures) or is currently on medication lowering seizure threshold (e.g. tricyclic antidepressants) or has used seizure threshold lowering medication within 14 days prior to administration of the preparation.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving adequate bowel cleansing based on Boston Bowel Preparation Scale (BBPS) | Day 2
  To describe the success rate of bowel cleansing in paediatric participants after administration of PLENVU® or sodium picosulfate as measured by the BBPS. The BBPS is a scoring system used to assess bowel cleanliness during colonoscopy. The scale ranges from 0 to 3, evaluating the three colonic segments (i.e. right colon, transverse colon, and left colon) where a score of 0 indicates an unprepared colon segment with mucosa not visible due to solid stool, and 3 indicates mucosa of colon segment seen well, with bowel cleansing success defined as a score of ≥2 in all three segments.

SECONDARY OUTCOMES:
Percentage of participants achieving successful bowel cleansing based on Harefield Cleansing Scale (HCS) | Day 2
  To describe the success rate of bowel cleansing in paediatric participants after administration of PLENVU® or sodium picosulfate as measured by the HCS. The HCS is scoring system used to assess bowel cleanliness during colonoscopy. The scale ranges from 0 to 4 evaluating five segments (i.e. ascending colon, transverse colon, descending colon, sigmoid colon and rectum). The scores of the five segments will be the basis for a final grading of A, B, C, or D. Success is defined as a HCS grade of A or B.
Number of participants with Adverse events (AEs) and Serious adverse events (SAEs) | From Screening (Day -28 to Day -1) to safety follow-up (Day 9 ± 2 days)
  To determine the safety of PLENVU® as compared to sodium picosulfate in paediatric participants.
Number of participants with a response on the Likert Scale | Day 1 and Day 2
  To determine the tolerability, palatability and acceptability of PLENVU® as compared to sodium picosulfate. A paediatric 5-point Likert Scale will be used to assess the tolerability, palatability and acceptability. It uses a combination of facial expressions and simple language to make it easier for children to understand and respond.

CONTACTS AND LOCATIONS:
Locations (40):
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem, Antwerp
  - Universitair Ziekenhuis Brussel (AZ-VUB - Academisch Ziekenhuis der Vrije Universiteit Brussel), Jette, Brussels Capital
  - Clinique CHC MontLegia, Alleur, Liege
- Germany (5):
  - Krankenhaus Barmherzige Brueder Regensburg - Klinik fuer Kinder- und Jugendmedizin, Regensburg, Bavaria
  - Universitaetsklinikum Muenster (UKM) - Klinik fuer Kinder- und Jugendmedizin - Allgemeine Paediatrie, Münster, North Rhine-Westphalia
  - Helios Uniklinikum Wuppertal, Wuppertal, North Rhine-Westphalia
  - Universitätsmedizin Der Johannes Gutenberg-Universität Mainz KöR, Mainz, Rhineland-Palatinate
  - Charité Universitätsmedizin Berlin, Berlin
- Hungary (3):
  - Semmelweis Egyetem Gyermekgyogyaszati Klinika Bokay Utcai Reszleg, Budapest
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet, Budapest
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktato Korhaz, Miskolc
- Italy (9):
  - Azienda Ospedaliera Universitaria Meyer IRCCS, Florence, Firenze
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria Gaetano Martino, Messina
  - Ospedale Maggiore Policlinico, Fondazione IRCCS Ca' Granda, Milan
  - Azienda Ospedaliera Universitaria Federico II - Pediatria Generale, Napoli
  - AOU Università degli studi della Campania Luigi Vanvitelli, Policlinico di Napoli - Pediatria, Napoli
  - Azienda Ospealiero Universitaria Policlinico Umberto I, Roma
  - Policlinico Gemelli - Endoscopia Digestiva Chirurgica, Roma
  - Azienda Ospedaliero-Universitaria Sant'Andrea - Pediatria, Roma
- Netherlands (3):
  - Amphia Hospital - Pediatrics, Breda, North Brabant
  - Amsterdam UMC - Pediatrics, Amsterdam, North Holland
  - Isala Klinieken, Zwolle, Overijssel
- Poland (6):
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu - Oddzial Pediatrii i Gastroenterologii, Torun, Kuyavian-Pomeranian Voivodeship
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow, Lesser Poland Voivodeship
  - Instytut "Pomnik - Centrum Zdrowia Dziecka" - Oddzial Gastroenterologii, Hepatologii, Zaburzen Odzywiania i Pediatrii, Warsaw, Masovian Voivodeship
  - Uniwersytecki Dzieciecy Szpital Kliniczny Imienia Ludwika Zamenhofa w Bialymstoku - Klinika Pediatrii, Gastroenterologii, Hepato, Bialystok, Podlaskie Voivodeship
  - Gdanski Uniwersytet Medyczny (GUMed) - Katedra i Klinika Pediatrii, Gastroenterologii, Alergologii i Zywienia Dzieci, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. prof. Stanislawa Szyszko SUM w Katowicach Oddzial Gastroenterologii i Hepatolog, Zabrze, Silesian Voivodeship
- Spain (5):
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Parc Tauli Hospital Universitarli, Sabadell, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Materno Infantil de Málaga, Málaga
- United Kingdom (6):
  - NHS Lothian - Royal Hospital for Children & Young People, Edinburgh, Edinburgh, City of
  - King's College Hospital NHS Foundation Trust, London, York
  - Birmingham Women's and Children's NHS Foundation Trust - Birmingham Children's Hospital, Birmingham
  - Barts Health NHS Trust, London
  - Great North Children's Hospital - Royal Victoria Infirmary, Newcastle upon Tyne
  - Sheffield Children's NHS Foundation Trust - Sheffield Children's Hospital, Sheffield